CLINICAL TRIAL: NCT05845853
Title: Effect of Scapular Motor Control Exercise in Patient With Chronic Mechanical Neck Pain
Brief Title: Scapular Motor Control for Chronic Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aisha Said ABDEL Raouf Agoor, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: motor control in neck pain
Record Dates: First submitted 2023-03-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Mechanical Neck Pain

STUDY DESIGN:
Intervention Model Description: This will be a double blinded, randomized, controlled, pre-post test clinical trial
Who Masked: Participant, Investigator
Masking Description: Patients will be randomly assigned into one of the two groups. We will use a simple randomization method to allocate participants to the groups. A random number generator available online from www.randomization.com will be used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventinal group (Experimental): 28 subject will receive a program of scapular motor control exercises using PNF technique in addition to the conventional treatment for 18 sessions (3 sessions per week for six weeks)
  Interventions: Other: scapular PNF technique
- control group (No Intervention): 28 subject will receive conventional physical therapy program (heat-TENS) for 18 sessions (3 sessions per week for six weeks)

INTERVENTIONS:
Other: scapular PNF technique — PNF Technique is based on movement patterns to facilitate and correct sensory-motor function,then correct the impaired impulses emerging from proprioceptive receptors in the muscle. Therefore, it decreases pain and improve the strength of muscles.
  PNF position renders a greater amount of sensory input coming from the periphery than that in the neutral position .
  Arms: interventinal group

SUMMARY:
The purpose of this study is to investigate the effect of motor control training using scapular PNF exercise on neck pain, function, proprioception, and scapular muscle strength in patients with chronic mechanical neck pain.

DETAILED DESCRIPTION:
Chronic mechanical neck pain (CMNP) is defined as generalized neck and/ or shoulder pain for more than 3 months with symptoms provoked by neck movement, neck postures, or palpation of the cervical muscles .

regional interdependence (RI) is defined as the concept that a patient's primary musculoskeletal symptom(s) may be directly or indirectly related or influenced by impairments from various body regions and systems regardless of proximity to the primary symptom(s)'.

Changes in scapular posture and alteration of muscle activation patterns of scapulothoracic muscles are cited as potential risk factors for neck pain the structural connectivity of the cervical spine and scaopulothorathic muscles . The bones and muscles of the cervical spine and the shoulders are connected to each other mechanically, thus a continuously applied mechanical load on the shoulders directly increases the load on the cervical region, which may cause joint and ligament pain Scapular malalignment can contribute to prolonged compressive loading of the posterior cervical structures .

It has been suggested that abnormal joint stress affects the firing of cervical afferents, leading to changes in proprioceptive function. Moreover, pain leads to changes in motor control . we believe that scapular motor control exercises using PNF technique may help to restore normal alignment and reverse this vicious circle PNF Technique is based on movement patterns to facilitate and correct sensory-motor function it has been suggested that PNF correct the impaired impulses emerging from proprioceptive receptors in the muscle. Therefore, it decreases pain and desires to improve the strength of muscles. PNF position renders a greater amount of sensory input coming from the periphery than that in the neutral position .The purpose of this study is to investigate the effect of motor control training using scapular PNF exercise on neck pain, function, proprioception, and scapular muscle strength in patients with chronic mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* -The subject will be referred from orthopedic surgeon with diagnosis of CMNP.
* Subjects with CMNP of more than 3 months with age range between 18 and 45 years
* Subjects having a baseline NDI score of at least 20% (10 points)
* At least 3/10 pain intensity on VAS

Exclusion Criteria:

* Spinal canal stenosis.
* Traumatic injury to the cervical spine.
* Previous surgery related to cervical spine.
* Hypermobility of the cervical spine,
* Any red flags e.g. cervical instability, history of cancer, long use of corticosteroids.
* Presence of an inflammatory rheumatologic disease,

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
change in cervical pain | one week after end of treatment
  by using the Arabic version of Numeric pain rating scale , ranging from 0 ("no pain") to 10 ("worst pain imaginable")
change in neck function | one week after end of treatment
  by using the Arabic version of neck disability index that consists of 10 questions: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 (no disability) to 5 (total disability). The maximum possible score is 50.
change in proprioceptive inputs of cervical | one week after end of treatment
  Bubble Inclinometer will be used to assess proprioceptive inputs of cervical
  * flexion - extension
  * right side bending - left side bending
  * cervical right rotate - cervical left rotation
change in muscle strength | one week after end of treatment
  Hand-held dynamometer will be used to assess muscle strength
  * upper trapezius - middle trapezius
  * lower trapezius - serratus anterior

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Tala Central Hospital, Tala, Munofia
  - Tala Central Hospital, Tala

REFERENCES:
- See also: Bansal, R., & Paul, M. (2020). Effectiveness of Motor Control Therapeutic Exercise Vs. Proprioceptive Neuromuscular Facilitation in Subjects With Cervical Spondylosis on Pain and Functional Disability. International Journal of Physiotherapy and Researc — https://doi.org/10.16965/ijpr.2020.162
- See also: Celenay, S. T., Kaya, D. O., & Akbayrak, T. (2016). Cervical and scapulothoracic stabilization exercises with and without connective tissue massage for chronic mechanical neck pain: A prospective, randomised controlled trial. Manual Therapy, 21, 144-150. — https://doi.org/10.1016/j.math.2015.07.003
- See also: Ha, S. min, Kwon, O. yun, Yi, C. hwi, Jeon, H. seon, & Lee, W. hwee. (2011). Effects of passive correction of scapular position on pain, proprioception, and range of motion in neck-pain patients with bilateral scapular downward-rotation syndrome. Manu — https://doi.org/10.1016/j.math.2011.05.011
- See also: 25. Ijspeert, J., Kerstens, H. C. J. W., Janssen, R. M. J., Geurts, A. C. H., Van Alfen, N., & Groothuis, J. T. (2019). Validity and reliability of serratus anterior hand held dynamometry. BMC Musculoskeletal Disorders, 20(1), 1-8. — https://doi.org/10.1186